CLINICAL TRIAL: NCT06782386
Title: A Prospective Observational Study Evaluating the Effectiveness of Photographic and Thermal Monitoring in the Management of High-risk Diabetic Foot Patients
Brief Title: Remote Temperature and Visual Monitoring To Help Manage Diabetic Foot Ulcers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bluedrop Medical Limited (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BMS CP003
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: DFU; Remote monitoring; Thermovisual monitoring
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Use of device (Active Comparator): This cohort will be recruited to use the OneStep Foot Scanner in their homes everyday for 12 months
  Interventions: Device: OneStep Foot Scanner
- Control Group from Retrospective Patient Database (No Intervention): Patients with a history of previous DFU(s) will be matched with participants in the active arm and analyzed

INTERVENTIONS:
Device: OneStep Foot Scanner — Daily scans with the OneStep Foot scanner will provide thermal and visual data of the soles of the feet to assist in early identification of risk factors associated with Diabetic Foot Ulcers
  Arms: Use of device

SUMMARY:
This study is a prospective, observational investigation evaluating the effectiveness of Remote ThermoVisual Monitoring (RTVM) in the early detection of diabetic foot ulcers (DFUs) in high-risk populations. The primary objective is to compare the incidence of Wagner stage 2 or higher DFUs at the time of presentation between patients using RTVM and a matched control group from a retrospective patient database.

Participants will include adults aged 18 years or older with type 1 or type 2 diabetes mellitus and a history of a plantar DFU that healed within the past five years. The study will enroll approximately 100 participants across up to 30 centers affiliated with SerenaGroup®. The intervention involves daily use of the OneStep Foot Scanner™, which measures temperature and captures visual images of the soles of the feet to detect signs of inflammation or anomalies.

Secondary objectives include evaluating ulcer-free survival, amputation-free survival, time to first evaluation for new DFUs, and healthcare utilization rates. Exploratory endpoints will assess neuropathy-specific quality of life and the costs associated with ulcer and amputation care. Participants will be monitored over a period of 12 months.

Results from this study aim to provide insights into the efficacy of RTVM as a preventative tool for managing diabetic foot health and reducing the burden of DFUs in high-risk populations.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, observational investigation designed to assess the utility of Remote ThermoVisual Monitoring (RTVM) using the OneStep Foot Scanner™ in detecting diabetic foot ulcers (DFUs) at an earlier stage in high-risk populations. DFUs represent a significant clinical and economic burden, often leading to severe complications, including infections and amputations. Early detection and intervention are critical to reducing morbidity and improving patient outcomes.

The primary objective is to compare the incidence of Wagner stage 2 or higher DFUs at the time of presentation in participants using RTVM to a matched historical control group. The secondary objectives include ulcer-free survival, amputation-free survival, time to first evaluation for new DFUs, and healthcare utilization rates. Exploratory endpoints include assessing neuropathy-specific quality of life and evaluating the economic impact of RTVM on DFU and amputation care costs.

The study will enroll approximately 100 participants aged 18 years or older with a confirmed diagnosis of type 1 or type 2 diabetes mellitus and a history of plantar DFUs that have healed within the past five years. Eligible participants will be recruited across up to 30 SerenaGroup® clinical sites. Participants will use the OneStep Foot Scanner™ daily to capture thermographic and visual data of the soles of their feet, which will be analyzed to identify signs of inflammation, potential ulceration, or other abnormalities. The data collected will be reviewed periodically by healthcare professionals for signs requiring intervention.

Participants will be followed for a period of 12 months, during which they will undergo regular clinical evaluations and remote monitoring assessments. The study will not only evaluate the effectiveness of RTVM in reducing the severity of DFUs but also explore its impact on healthcare costs, quality of life, and overall disease management strategies.

This study aims to provide critical insights into the feasibility of implementing RTVM as a preventive tool in routine diabetic foot care and its potential role in mitigating the global burden of DFUs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Diagnosis of type 1 or type 2 diabetes mellitus
* History of a plantar DFU within 5 years of enrollment.
* Access to a phone on which they can receive study communications.
* SUBGROUP: a patient with an active Wagner grade 1 DFU may be enrolled if in the opinion of the investigator the wound is sufficiently epithelialized and can withstand the pressure applied during scanning.

Exclusion Criteria:

* Weight, when fully clothed, of greater than 300 kg (~330 lbs) NOTE: for participants over 150kg the device will need to be used from a seated position
* Active Charcot arthropathy defined as the phase where the foot is undergoing collapse
* Active foot infection or gangrene
* Critical limb threatening ischemia as evidenced by rest pain, or the presence of gangrene on any part of the foot.
* Any mental health disorder, psychiatric disorder, or alcohol or drug abuse history such that, in the opinion of the investigator, rule the patient is unreliable as a study participant
* Any travel plans expected to result in an interruption of device use for greater than 30 consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of more severe DFUs presenting | 12 months
  Incidence of Wagner grade 2 or higher ulcer at the time of first presentation for patients with a history of DFUs that healed in the previous 5 years.

SECONDARY OUTCOMES:
Length of time to DFU development | 12 months
  Time to first evaluation in patients with new DFUs in a high-risk population of patients with healed (within 5 years) DFUs
Number of Patients who Experience Ulcer Free Survival | 12 months
  Ulcer free survival (of Wagner Grade 2 or higher ulcers), in a high-risk population of patients with recently healed DFUs.
Number of Patients who Experience Amputation Free Survival | 12 months
  Amputation free survival in a high-risk population of patients with recently healed DFUs
Resource utilization | 12 months
  Incidence of inpatient admissions, emergency room visits and outpatient provider encounters in patients with new DFUs in a high-risk population of patients with recently healed DFUs
Compliance with Recommended Device Use as Measured by Scan Data Collected from the Bluedrop OneStep Foot Scanner | 12 months
  Adherence with RTVM in participants assigned to use RTVM

OTHER OUTCOMES:
PROM | 12 months
  Survey-ascertained participant reported quality of life measures using the NEUROPATHY-SPECIFIC QUALITY OF LIFE Questionnaire using a Likert scale of 1 to 5 for frequency of symptoms where 1 represents "never" and 5 represents "all the time" - with higher scores signifying a poorer quality of life.
Resource utilization costs | 12 months
  Costs associated with ulcer and amputation care in a high-risk population of patients with recently healed DFUs

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, Principal Investigator — Serena Group
Locations (2):
- United States (2):
  - Three Rivers Wound and Hyperbaric Center, North Port, Florida
  - SerenaGroup Monroeville, Monroeville, Pennsylvania